CLINICAL TRIAL: NCT02776033
Title: A Multicentre, Randomised, Double-blind (Sponsor-unblinded), Placebo-controlled, Repeat Dose Study to Investigate the Safety and Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of GSK2982772 in Subjects With Active Plaque-type Psoriasis
Brief Title: Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of Repeat Doses of GSK2982772 in Subjects With Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 203167
Record Dates: First submitted 2016-05-16; First posted 2016-05-18 (Estimated); Results first posted 2019-08-22 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-06

CONDITIONS: Psoriasis
Keywords: tolerability; safety; GSK2982772; RIP1 kinase inhibitor; psoriasis
MeSH Terms: conditions — Psoriasis | interventions — GSK2982772

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- GSK2982772 receivers in Cohort 1 (Experimental): Randomized subjects will receive GSK2982772 BID (approximately 12 hours apart) via oral route for 84 days.
  Interventions: Drug: GSK2982772
- Placebo receivers in Cohort 1 (Placebo Comparator): Randomized subjects will receive placebo BID via oral route for 84 days.
  Interventions: Drug: Placebo
- GSK2982772 receivers in Cohort 2 (Experimental): Randomized subjects will receive GSK2982772 TID (approximately 8 hours apart) via oral route for 84 days
  Interventions: Drug: GSK2982772
- Placebo receivers in Cohort 2 (Placebo Comparator): Randomized subjects will receive placebo TID via oral route for 84 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK2982772 — GSK2982772 will be supplied as a white to almost white, round, film coated 30 mg oral tablets; two tablets to be taken in the morning and two in the evening, as directed for Cohort 1 and for Cohort 2 two tablets to be taken three times daily as directed.
  Arms: GSK2982772 receivers in Cohort 1; GSK2982772 receivers in Cohort 2
Drug: Placebo — Matching placebo will be supplied as a white to almost white, round film coated tablets; two tablets to be taken in the morning and two in the evening, as directed for Cohort 1 and for Cohort 2 two tablets to be taken three times daily as directed.
  Arms: Placebo receivers in Cohort 1; Placebo receivers in Cohort 2

SUMMARY:
This is the first study with GSK2982772, a receptor-interacting protein-1 (RIP1) kinase inhibitor, in subjects with active plaque-type psoriasis (PsO). The primary objective will be to investigate the safety and tolerability of repeat oral doses of GSK2982772 60 milligram (mg) twice daily (BID) for 84 days in Cohort 1 and 60 mg thrice daily (TID) for 84 days in Cohort 2. In addition, a number of experimental and clinical endpoints will be employed to obtain information on the pharmacokinetics, pharmacodynamics, and efficacy in subjects with active PsO. There will be two Cohorts of subjects. In Cohort 1 after a screening period of up to 30 days, approximately 30 subjects will be randomized to receive either GSK2982772 60 mg BID or placebo for 84 days (12 Weeks), followed by a follow-up period (28 days). In Cohort 2 after a screening period of up to 30 days, approximately 24 subjects will be randomized to receive either GSK2982772 60 mg TID or placebo for 84 days (12 Weeks), followed by a follow-up period (28 days). The total duration of participation is approximately 20 Weeks from screening to the last study visit.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 75 years of age inclusive, at the time of signing the informed consent.
* Subjects who do not have any medical conditions, other than active plaque-type psoriasis, that in the opinion of the Investigator put the subject at unacceptable risk or interfere with study assessments or integrity of the data. All medical conditions must be stable for the duration of the study.
* Presence of active chronic plaque-type psoriasis as determined by the Investigator for at least 6 months (confirmed by the subject or medical record) before first dose of study treatment (Day 1).
* Subject has psoriasis plaques involving Body Surface Area >=3% assessed at screening and before dosing on Day 1.
* Physician Global Assessment >=3.
* Subject must agree to avoid prolonged exposure to natural sunlight, tanning beds or phototherapy devices for the duration of the study
* Subject has at least two stable plaques assessed at screening and before dosing on Day 1:

Both must be of a suitable size (>=3 centimeter [cm] by 3 cm) and one in a site suitable for repeat biopsy, and one in a site suitable for index lesion PLSS scoring.

Both plaques must have a PLSS lesional score >=2 for the induration component (moderate or above), >=1 for erythema and scaling with a total score of >=5.

The biopsy lesion must not be on the face, groin, scalp, knees, elbows, or on the palmar/plantar surfaces of the hands/feet, and must be shielded from natural light with clothing.

* Subject is naive to any biologic therapies for psoriasis, OR has had previous exposure to a single anti- TNF biologic agent in the context of a previous clinical trial. The anti-TNF biologic agent must have been discontinued more than 8 weeks prior to screening visit (12 Weeks or 5 half lives whichever is longer from first dose).
* A body mass index within the range of 18.5-35 kilogram per meter square (kg)/m^2 (inclusive).
* Male and Female subjects:

Males: Male subjects with female partners of child bearing potential must comply with the pre specified contraception requirements.

Females: A female subject is eligible to participate if she is not pregnant (as confirmed by a negative serum or urine human chorionic gonadotropin test), not lactating, and is either of non-reproductive potential or reproductive potential. If of reproductive potential, then the subject should agree to follow one of the options listed per GSK Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential from 30 days prior to the first dose and until 30 days after the last dose of study medication The Investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.

* Capable of giving signed informed consent

Exclusion Criteria:

* Subjects with clinically overt concurrent psoriatic arthritis who are receiving chronic disease-modifying anti-rheumatic medications therapy (other than non-steroidal anti-inflammatory drug), as judged by the Investigator.
* Has nonplaque forms of psoriasis (e.g. erythrodermic, guttate, or pustular), as judged by the Investigator.
* Has current drug-induced psoriasis (e.g., a new onset of psoriasis or an exacerbation from beta blockers, calcium channel blockers, or lithium).
* Subject with current history of Suicidal Ideation Behaviour as measured using the Columbia Suicide Severity Rating Scale or a history of attempted suicide.
* An active infection, or a history of infections as follows:

Hospitalization for treatment of infection within 60 days before first dose (Day 1).

Currently on any suppressive therapy for a chronic infection (such as pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster and atypical mycobacteria).

Use of parenteral (intravenous or intramuscular) antibiotics (antibacterials, antivirals, antifungals, or antiparasitic agents) within 60 days before first dose.

A history of opportunistic infections within 1 year of screening (e.g. pneumocystis jirovecii, cytomegalovirus, pneumonitis, aspergillosis). This does not include infections that may occur in immunocompetent individuals, such as fungal nail infections or vaginal candidiasis, unless it is of an unusual severity or recurrent nature.

Recurrent or chronic infection or other active infection that, in the opinion of the Investigator might cause this study to be detrimental to the subject.

History of tuberculosis (TB), irrespective of treatment status. A positive diagnostic TB test at screening defined as a positive QuantiFERON-TB Gold test or T-spot test.

In cases where the QuantiFERON or T-spot test is indeterminate, the subject may have the test repeated once, but they will not be eligible for the study unless the second test is negative.

In cases where the QuantiFERON or T-spot test is positive, but a locally-read follow up chest X-ray, shows no evidence of current or previous pulmonary tuberculosis, the subject may be eligible for the study at the discretion of the Investigator and medical monitor.

* ECG for heart rate QTc >450 milliseconds (msec) or QTc >480 msec in subjects with bundle branch block.
* Alanine aminotransferase >2×upper limit of normal (ULN) and bilirubin >1.5×ULN (isolated bilirubin >1.5×ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%) at screening.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Current or history of renal disease or estimated glomerular filtrate rate by Chronic Kidney Disease Epidemiology Collaboration equation <60 mL/min/1.73 m^2.
* Hereditary or acquired immunodeficiency disorder, including immunoglobulin deficiency.
* A major organ transplant (e.g., heart, lung, kidney, liver) or hematopoietic stem cell/marrow transplant.
* A planned surgical procedure that, in the opinion of the Investigator, makes the subject unsuitable for the study.
* A history of malignant neoplasm within the last 5 years, except for adequately treated cancers of the skin (basal or squamous cell carcinoma) or carcinoma in situ of the uterine cervix that has been fully treated and shows no evidence of recurrence.
* A history of hypertrophic scarring or keloid formation, or known allergy to lidocaine or other local anaesthetics.
* The subject has received treatment with the specified therapies listed in the protocol, or changes to those treatments, within the specified timeframe.

Other medications (including vitamins, herbal and dietary supplements) will be considered on a case-by-case basis, and will be allowed if in the opinion of the Investigator the medication will not interfere with the study procedures or compromise subject safety.

* History of alcohol or drug abuse that would interfere with the ability to comply with the study.
* Subject intends to sunbathe or use a tanning device (sun bed or solarium) within 14 days prior to Day 1 and until completion of the follow up visit (Day 112).
* History of sensitivity to any of the study treatments, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicates their participation.
* Received a live or attenuated vaccine within 30 days of randomization OR plan to receive a vaccination during the study until completion of the follow-up visit.
* The subject has participated in a clinical trial and has received an investigational product within 30 days or 5 half-lives, whichever is longer before the first dose of study medication, or plans to take part in another clinical trial at the same time as participating in this clinical trial. Subjects who were randomized into Cohort 1 are not eligible to be re-randomized into Cohort 2.
* Hemoglobin <11 g/deciliter (dL); hematocrit <30%, white blood cell count =<3,000/millimeter (mm)^3 (<=3.0×10^9/L) ; platelet count <=100,000/microliter (µL) (<=100 × 10^9/L); absolute neutrophil count <=1.5×10^9/L at the screening visit.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment. As potential for and magnitude of immunosuppression with this compound is unknown, subjects with presence of hepatitis B core antibody (HBcAb) should be excluded. Subjects positive for HBsAg and/or positive for anti-HBcAb (regardless of anti-HBs antibody status) are excluded.
* A positive serology for human immunodeficiency virus 1 or 2 at screening.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 3 months.
* Exposure to more than 4 investigational medicinal products within 12 months prior to the first dosing day

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-08-30 (Actual); Primary Completion 2018-01-04 (Actual); Study Completion 2018-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Canada (4):
  - GSK Investigational Site, Markham, Ontario
  - GSK Investigational Site, Peterborough, Ontario
  - GSK Investigational Site, Waterloo, Ontario
  - GSK Investigational Site, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20374

REFERENCES:
- [Background] Weisel K, Berger S, Papp K, Maari C, Krueger JG, Scott N, Tompson D, Wang S, Simeoni M, Bertin J, Peter Tak P. Response to Inhibition of Receptor-Interacting Protein Kinase 1 (RIPK1) in Active Plaque Psoriasis: A Randomized Placebo-Controlled Study. Clin Pharmacol Ther. 2020 Oct;108(4):808-816. doi: 10.1002/cpt.1852. Epub 2020 Jul 7. PMID 32301501

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a repeat dose study in participants with active plaque-type psoriasis. Participants received either GSK2982772 60 milligrams (mg) or placebo orally twice daily (BID) in Cohort 1 and either GSK2982772 60 mg or placebo orally three times daily (TID) in Cohort 2. The study was conducted at 4 centers in Canada.
Pre-assignment Details: A total of 100 participants were screened, of which, 65 participants were enrolled in the study.
Groups:
- Placebo: Eligible participants received placebo orally BID, for 12 weeks in Cohort 1 and orally TID for 12 weeks in Cohort 2 of the study.
- GSK2982772 60 mg BID: Eligible participants received GSK2982772, 60 mg orally BID for 12 weeks in Cohort 1 of the study.
- GSK2982772 60 mg TID: Eligible participants received GSK2982772, 60 mg orally TID for 12 weeks in Cohort 2 of the study.
Period: Overall Study
Arm/Group | Placebo | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Started | 18 | 23 | 24
Completed | 14 | 21 | 22
Not Completed | 4 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 2
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Adverse Event | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK2982772 60 mg BID | GSK2982772 60 mg TID | Total
Number analyzed (Participants) | 18 | 23 | 24 | 65
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.1 (14.95) | 44.6 (12.52) | 47.5 (13.41) | 46.3 (13.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 5 | 16
  Male | 13 | 17 | 19 | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - Central/South Asian Heritage | 2 | 1 | 2 | 5
  Asian - East Asian Heritage | 1 | 1 | 0 | 2
  Asian - South East Asian Heritage | 1 | 1 | 1 | 3
  Native Hawaiian or other Pacific Islander | 0 | 0 | 1 | 1
  White - Arabic/North African Heritage | 1 | 1 | 1 | 3
  White - White/Caucasian/European Heritage | 13 | 19 | 19 | 51

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Non-SAEs
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, is associated with liver injury and impaired liver function or any other situations as per medical or scientific judgment. Safety Population comprised of all participants who received at least one dose of study treatment.
Time Frame: Up to Day 116
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 18 | 23 | 24
Participants
  Any SAE | 0 | 1 | 1
  Any non-SAE | 8 | 21 | 16

2. Primary Outcome: Number of Participants With Worst-case Post-Baseline Clinical Chemistry Results by Potential Clinical Importance (PCI) Criteria
Description: Blood samples were collected for analysis of clinical chemistry parameters. Clinical concern ranges were >=2x Upper Limit of Normal (ULN) units per liter (U/L) for alanine aminotransferase (ALT), <30 millimoles per liter (mmol/L) for albumin, >=2x ULN U/L for alkaline phosphatase, >=2x ULN U/L for aspartate aminotransferase (AST), <2 or >2.75 mmol/L for Calcium, >44.2 mmol/L for Creatinine, <3 or >9 mmol/L for Glucose, <3 or>5.5 mmol/L for Potassium, <130 or >150 mmol/L for Sodium, and >=1.5xULN micromoles per liter for total bilirubin. Participants were counted in worst case category that their value changes to (Low, Normal or High), unless there is no change in their category. Participants whose value category was unchanged (example given [e.g.], High to High), or whose value became normal, were recorded in "To Normal or No Change" category. Participants were counted twice if they had values that changed 'To Low' and 'To High', Baseline is defined as the latest pre-dose assessment.
Time Frame: Up to Day 116
Population: Safety Population. Only those clinical chemistry parameters with data available per PCI criteria have been presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 18 | 23 | 24
Participants
  ALT; To Low | 0 | 0 | 0
  ALT; To Normal or No Change | 18 | 22 | 24
  ALT; To High | 0 | 1 | 0
  Albumin; To Low | 0 | 0 | 0
  Albumin; To Normal or No Change | 18 | 23 | 24
  Albumin; To High | 0 | 0 | 0
  Alkaline phosphatase; To Low | 0 | 0 | 0
  Alkaline phosphatase; To Normal or No Change | 18 | 23 | 24
  Alkaline phosphatase; To High | 0 | 0 | 0
  AST; To Low | 0 | 0 | 0
  AST; To Normal or No Change | 18 | 23 | 24
  AST; To High | 0 | 0 | 0
  Calcium; To Low | 0 | 0 | 0
  Calcium; To Normal or No Change | 18 | 23 | 24
  Calcium; To High | 0 | 0 | 0
  Creatinine; To Low | 0 | 0 | 0
  Creatinine; To Normal or No Change | 18 | 21 | 24
  Creatinine; To High | 0 | 2 | 0
  Glucose; To Low | 0 | 1 | 0
  Glucose; To Normal or No Change | 16 | 22 | 23
  Glucose; To High | 2 | 1 | 1
  Potassium; To Low | 0 | 0 | 0
  Potassium; To Normal or No Change | 18 | 22 | 24
  Potassium; To High | 0 | 1 | 0
  Sodium; To Low | 0 | 0 | 0
  Sodium; To Normal or No Change | 18 | 23 | 24
  Sodium; To High | 0 | 0 | 0
  Total bilirubin; To Low | 0 | 0 | 0
  Total bilirubin; To Normal or No Change | 17 | 23 | 24
  Total bilirubin; To High | 1 | 0 | 0

3. Primary Outcome: Number of Participants With Worst-case Post-Baseline Hematology Results by PCI Criteria
Description: Blood samples were collected for analysis of hematology parameters. Clinical concern ranges were >0.54 calculated as proportion of red blood cells in blood for Hematocrit, >180 grams per liter for Hemoglobin, <0.8 x10^9 cells per liter for Lymphocytes, <1.5 x10^9 cells per liter for Neutrophil count, <100 or >550 x10^9 cells per liter for Platelet count and <3 or >20 x10^9 cells per liter White Blood Cell count. Participants were counted in the worst case category that their value changes to (Low, Normal or High), unless there is no change in their category. Participants whose value category was unchanged (e.g., High to High), or whose value became normal, are recorded in the "To Normal or No Change" category. Participants were counted twice if they had values that changed 'To Low' and 'To High'. Baseline is defined as the latest pre-dose assessment.
Time Frame: Up to Day 116
Population: Safety Population. Only those hematology parameters with data available per PCI criteria have been presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 18 | 23 | 24
Participants
  Hematocrit; To Low | 0 | 0 | 0
  Hematocrit; To Normal or No Change | 18 | 23 | 22
  Hematocrit; To High | 0 | 0 | 2
  Hemoglobin; To Low | 0 | 0 | 0
  Hemoglobin; To Normal or No Change | 17 | 23 | 23
  Hemoglobin; To High | 1 | 0 | 1
  Lymphocytes; To Low | 1 | 1 | 0
  Lymphocytes; To Normal or No Change | 17 | 22 | 24
  Lymphocytes; To High | 0 | 0 | 0
  Neutrophil count; To Low | 0 | 0 | 0
  Neutrophil count; To Normal or No Change | 18 | 23 | 24
  Neutrophil count; To High | 0 | 0 | 0
  Platelet count; To Low | 0 | 0 | 0
  Platelet count; To Normal or No Change | 18 | 23 | 24
  Platelet count; To High | 0 | 0 | 0
  White Blood Cell count; To Low | 0 | 0 | 0
  White Blood Cell count; To Normal or No Change | 18 | 23 | 24
  White Blood Cell count; To High | 0 | 0 | 0

4. Primary Outcome: Change From Baseline in Urine Potential of Hydrogen (pH)
Description: Urine samples were collected for measurement of urine pH at indicated time points. pH is a measure of hydrogen ion concentration and used to determine the acidity or alkalinity of urine. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Baseline is defined as the latest pre-dose assessment. Change from Baseline is defined as any post-dose visit value minus Baseline value.
Time Frame: Baseline (Pre-dose on Day 1), Day 8, Day 15, Day 43, Day 85 and Follow-up (Day 116)
Population: Safety Population. Only those participants with data available at specified time points were analyzed (represented by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Potential of hydrogen (pH)
Arm/Group | Placebo | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 18 | 23 | 24
Potential of hydrogen (pH)
  DAY 8; n=18, 23, 22: number analyzed (Participants) | 18 | 23 | 22
  DAY 8; n=18, 23, 22 | 0.69 (0.788) | -0.02 (0.730) | -0.11 (0.786)
  DAY 15; n=17, 21, 22: number analyzed (Participants) | 17 | 21 | 22
  DAY 15; n=17, 21, 22 | 0.56 (0.609) | 0.14 (0.673) | -0.16 (0.956)
  DAY 43; n=16, 21, 21: number analyzed (Participants) | 16 | 21 | 21
  DAY 43; n=16, 21, 21 | 0.22 (0.547) | 0.14 (0.655) | -0.36 (1.108)
  DAY 85; n=14, 21, 22: number analyzed (Participants) | 14 | 21 | 22
  DAY 85; n=14, 21, 22 | 0.29 (0.975) | 0.00 (0.592) | -0.32 (0.933)
  FOLLOW UP (Day 116); n=16, 22, 24: number analyzed (Participants) | 16 | 22 | 24
  FOLLOW UP (Day 116); n=16, 22, 24 | 0.25 (0.894) | -0.07 (0.541) | -0.17 (1.029)

5. Primary Outcome: Change From Baseline in Urine Specific Gravity
Description: Urine samples were collected to analyze specific gravity of urine. Specific gravity, is a measure of urine concentration and is measured using a chemical test. Specific gravity measurements provide a comparison of the amount of substances dissolved in urine as compared to pure water. If there were no solutes present, the specific gravity of urine would be 1.000 the same as pure water. Specific gravity between 1.002 and 1.035 could be considered as normal. Baseline is defined as the latest pre-dose assessment. Change from Baseline is defined as any post-dose visit value minus Baseline value.
Time Frame: Baseline (Pre-dose on Day 1), Day 8, Day 15, Day 43, Day 85 and Follow-up (Day 116)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 18 | 23 | 24
Ratio
  DAY 8; n=18, 23, 22: number analyzed (Participants) | 18 | 23 | 22
  DAY 8; n=18, 23, 22 | -0.0043 (0.00765) | -0.0020 (0.00704) | 0.0014 (0.00702)
  DAY 15; n=17, 21, 22: number analyzed (Participants) | 17 | 21 | 22
  DAY 15; n=17, 21, 22 | -0.0029 (0.00679) | -0.0028 (0.00567) | 0.0022 (0.00706)
  DAY 43; n=16, 21, 21: number analyzed (Participants) | 16 | 21 | 21
  DAY 43; n=16, 21, 21 | -0.0032 (0.00692) | 0.0000 (0.00649) | 0.0001 (0.00694)
  DAY 85; n=14, 21, 22: number analyzed (Participants) | 14 | 21 | 22
  DAY 85; n=14, 21, 22 | 0.0004 (0.00560) | -0.0022 (0.00608) | 0.0022 (0.00922)
  FOLLOW UP (Day 116); n=16, 22, 24: number analyzed (Participants) | 16 | 22 | 24
  FOLLOW UP (Day 116); n=16, 22, 24 | -0.0016 (0.00719) | -0.0020 (0.00739) | 0.0032 (0.00798)

6. Primary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Blood pressure was measured at indicated time points in supine or semi-supine position after 5 minutes rest. Baseline is defined as the latest pre-dose assessment. Change from Baseline is defined as any post-dose visit value minus Baseline value.
Time Frame: Baseline (Pre-dose on Day 1), Day 8, Day 15, Day 29, Day 43, Day 57, Day 71, Day 85 and Follow-up (Day 116)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Millimeter of mercury
Arm/Group | Placebo | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 18 | 23 | 24
Millimeter of mercury
  SBP; DAY 8; n=18, 23, 24 | 4.5 (12.27) | 4.7 (8.03) | 2.9 (12.19)
  SBP; DAY 15; n=17, 22, 24: number analyzed (Participants) | 17 | 22 | 24
  SBP; DAY 15; n=17, 22, 24 | 2.0 (10.55) | -1.0 (8.91) | -1.0 (7.96)
  SBP; DAY 29; n=16, 22, 24: number analyzed (Participants) | 16 | 22 | 24
  SBP; DAY 29; n=16, 22, 24 | 1.3 (11.52) | 3.3 (9.94) | -1.3 (13.26)
  SBP; DAY 43; n=16, 21, 23: number analyzed (Participants) | 16 | 21 | 23
  SBP; DAY 43; n=16, 21, 23 | -0.4 (14.65) | 0.1 (6.72) | -2.2 (10.51)
  SBP; DAY 57; n=14, 21, 22: number analyzed (Participants) | 14 | 21 | 22
  SBP; DAY 57; n=14, 21, 22 | -0.3 (12.63) | 2.6 (8.73) | 3.4 (15.70)
  SBP; DAY 71; n=14, 21, 22: number analyzed (Participants) | 14 | 21 | 22
  SBP; DAY 71; n=14, 21, 22 | 5.9 (15.08) | 2.5 (10.02) | -1.0 (12.95)
  SBP; DAY 85; n=14, 21, 22: number analyzed (Participants) | 14 | 21 | 22
  SBP; DAY 85; n=14, 21, 22 | 4.4 (10.36) | 2.9 (9.52) | -1.4 (10.93)
  SBP; FOLLOW UP (Day 116); n=16, 22, 24: number analyzed (Participants) | 16 | 22 | 24
  SBP; FOLLOW UP (Day 116); n=16, 22, 24 | 2.3 (14.64) | 2.7 (9.81) | 2.5 (13.61)
  DBP; DAY 8; n=18, 23, 24 | -0.4 (10.07) | 0.0 (5.72) | 1.4 (6.88)
  DBP; DAY 15; n=17, 22, 24: number analyzed (Participants) | 17 | 22 | 24
  DBP; DAY 15; n=17, 22, 24 | -1.5 (8.46) | -0.5 (6.68) | -2.3 (6.39)
  DBP; DAY 29; n=16, 22, 24: number analyzed (Participants) | 16 | 22 | 24
  DBP; DAY 29; n=16, 22, 24 | -1.4 (8.52) | -1.4 (7.75) | -1.2 (7.92)
  DBP; DAY 43; n=16, 21, 23: number analyzed (Participants) | 16 | 21 | 23
  DBP; DAY 43; n=16, 21, 23 | -0.6 (9.51) | 0.1 (6.69) | -1.8 (6.10)
  DBP; DAY 57; n=14, 21, 22: number analyzed (Participants) | 14 | 21 | 22
  DBP; DAY 57; n=14, 21, 22 | -2.4 (10.16) | 1.1 (6.09) | 2.0 (9.00)
  DBP; DAY 71; n=14, 21, 22: number analyzed (Participants) | 14 | 21 | 22
  DBP; DAY 71; n=14, 21, 22 | 1.1 (11.68) | -1.3 (8.12) | -0.8 (7.51)
  DBP; DAY 85; n=14, 21, 22: number analyzed (Participants) | 14 | 21 | 22
  DBP; DAY 85; n=14, 21, 22 | -0.6 (7.44) | -1.1 (4.54) | 0.1 (6.93)
  DBP; FOLLOW UP (Day 116); n=16, 22, 24: number analyzed (Participants) | 16 | 22 | 24
  DBP; FOLLOW UP (Day 116); n=16, 22, 24 | 0.9 (10.28) | 1.3 (7.40) | 1.3 (8.66)

7. Primary Outcome: Change From Baseline in Heart Rate
Description: Heart rate was measured at indicated time points in supine or semi-supine position after 5 minutes rest. Baseline is defined as the latest pre-dose assessment. Change from Baseline is defined as any post-dose visit value minus Baseline value.
Time Frame: Baseline (Pre-dose on Day 1), Day 8, Day 15, Day 29, Day 43, Day 57, Day 71, Day 85 and Follow-up (Day 116)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 18 | 23 | 24
Beats per minute
  DAY 8; n=18, 23, 24 | 2.8 (7.72) | 4.9 (10.54) | 2.3 (13.18)
  DAY 15; n=17, 22, 24: number analyzed (Participants) | 17 | 22 | 24
  DAY 15; n=17, 22, 24 | 1.5 (10.61) | 0.8 (8.43) | 1.9 (12.37)
  DAY 29; n=16, 22, 24: number analyzed (Participants) | 16 | 22 | 24
  DAY 29; n=16, 22, 24 | 1.0 (7.43) | 0.7 (9.61) | 4.0 (12.55)
  DAY 43; n=16, 21, 23: number analyzed (Participants) | 16 | 21 | 23
  DAY 43; n=16, 21, 23 | 0.2 (6.68) | 0.5 (7.64) | 4.9 (11.56)
  DAY 57; n=14, 21, 22: number analyzed (Participants) | 14 | 21 | 22
  DAY 57; n=14, 21, 22 | 2.9 (10.55) | 2.9 (10.42) | 5.3 (12.13)
  DAY 71; n=14, 21, 22: number analyzed (Participants) | 14 | 21 | 22
  DAY 71; n=14, 21, 22 | 1.6 (7.94) | 2.1 (8.81) | 2.4 (10.75)
  DAY 85; n=14, 21, 22: number analyzed (Participants) | 14 | 21 | 22
  DAY 85; n=14, 21, 22 | 0.9 (7.98) | 0.7 (8.63) | 1.9 (12.82)
  FOLLOW UP (Day 116); n=16, 22, 24: number analyzed (Participants) | 16 | 22 | 24
  FOLLOW UP (Day 116); n=16, 22, 24 | 3.5 (7.60) | 1.6 (10.28) | 5.1 (13.58)

8. Primary Outcome: Change From Baseline in Respiratory Rate
Description: Respiratory rate was measured at indicated time points in supine or semi-supine position after 5 minutes rest. Baseline is defined as the latest pre-dose assessment. Change from Baseline is defined as any post-dose visit value minus Baseline value.
Time Frame: Baseline (Pre-dose on Day 1), Day 8, Day 15, Day 29, Day 43, Day 57, Day 71, Day 85 and Follow-up (Day 116)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Placebo | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 18 | 23 | 24
Breaths per minute
  DAY 8; n=18, 23, 24 | -0.8 (2.18) | -0.4 (2.81) | 0.3 (2.86)
  DAY 15; n=17, 22, 24: number analyzed (Participants) | 17 | 22 | 24
  DAY 15; n=17, 22, 24 | 0.2 (3.21) | -0.6 (2.44) | -0.5 (2.45)
  DAY 29; n=16, 22, 24: number analyzed (Participants) | 16 | 22 | 24
  DAY 29; n=16, 22, 24 | 0.9 (3.34) | -0.8 (3.38) | 0.0 (4.01)
  DAY 43; n=16, 21, 23: number analyzed (Participants) | 16 | 21 | 23
  DAY 43; n=16, 21, 23 | -0.5 (2.68) | -0.4 (3.06) | 0.3 (3.50)
  DAY 57; n=14, 21, 22: number analyzed (Participants) | 14 | 21 | 22
  DAY 57; n=14, 21, 22 | 0.3 (3.12) | -0.5 (2.36) | -0.3 (3.08)
  DAY 71; n=14, 21, 22: number analyzed (Participants) | 14 | 21 | 22
  DAY 71; n=14, 21, 22 | 0.2 (3.09) | -0.5 (2.29) | 0.4 (3.53)
  DAY 85; n=14, 21, 22: number analyzed (Participants) | 14 | 21 | 22
  DAY 85; n=14, 21, 22 | 0.3 (3.31) | -0.5 (2.89) | -0.3 (3.76)
  FOLLOW UP (Day 116); n=16, 22, 24: number analyzed (Participants) | 16 | 22 | 24
  FOLLOW UP (Day 116); n=16, 22, 24 | 0.3 (1.62) | -0.1 (2.60) | -1.0 (3.22)

9. Primary Outcome: Change From Baseline in Body Temperature
Description: Body temperature was measured at indicated time points in supine or semi-supine position after 5 minutes rest. Baseline is defined as the latest pre-dose assessment. Change from Baseline is defined as any post-dose visit value minus Baseline value.
Time Frame: Baseline (Pre-dose on Day 1), Day 8, Day 15, Day 29, Day 43, Day 57, Day 71, Day 85 and Follow-up (Day 116)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Placebo | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 18 | 23 | 24
Celsius
  DAY 8; n=18, 23, 24 | 0.12 (0.544) | -0.11 (0.365) | 0.03 (0.656)
  DAY 15; n=17, 22, 24: number analyzed (Participants) | 17 | 22 | 24
  DAY 15; n=17, 22, 24 | 0.09 (0.466) | -0.04 (0.358) | 0.17 (0.538)
  DAY 29; n=16, 22, 24: number analyzed (Participants) | 16 | 22 | 24
  DAY 29; n=16, 22, 24 | -0.07 (0.447) | -0.03 (0.387) | 0.01 (0.749)
  DAY 43; n=16, 21, 23: number analyzed (Participants) | 16 | 21 | 23
  DAY 43; n=16, 21, 23 | -0.14 (0.358) | -0.01 (0.355) | 0.19 (0.757)
  DAY 57; n=14, 21, 22: number analyzed (Participants) | 14 | 21 | 22
  DAY 57; n=14, 21, 22 | 0.07 (0.705) | 0.11 (0.351) | 0.20 (0.646)
  DAY 71; n=14, 21, 22: number analyzed (Participants) | 14 | 21 | 22
  DAY 71; n=14, 21, 22 | -0.01 (0.487) | -0.17 (0.423) | -0.07 (0.667)
  DAY 85; n=14, 21, 22: number analyzed (Participants) | 14 | 21 | 22
  DAY 85; n=14, 21, 22 | 0.06 (0.483) | -0.03 (0.327) | 0.03 (0.562)
  FOLLOW UP (Day 116); n=16, 22, 24: number analyzed (Participants) | 16 | 22 | 24
  FOLLOW UP (Day 116); n=16, 22, 24 | -0.05 (0.459) | 0.02 (0.505) | 0.07 (0.624)

10. Primary Outcome: Number of Participants With Any Time Post-Baseline Results for Electrocardiogram Findings
Description: Single 12-lead electrocardiograms were obtained at indicated time points during the study using an electrocardiogram machine that automatically calculates the heart rate and measures PR, QRS, QT, QT interval corrected for heart rate (QTc) using Bazett's formula (QTcB) intervals and QTc using Fridericia's formula (QTcF). The abnormal findings were categorized as clinically significant (CS) and not clinically significant (NCS). Baseline is defined as the latest pre-dose assessment. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. The number of participants with normal and abnormal electrocardiogram findings at any time post-Baseline visit has been presented.
Time Frame: Up to Day 116
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 18 | 23 | 24
Participants
  Normal | 7 | 8 | 7
  Abnormal-NCS | 11 | 15 | 17
  Abnormal-CS | 0 | 0 | 0

11. Secondary Outcome: Plasma Concentrations of GSK2982772 at Days 43 and 85
Description: Blood samples were collected for pharmacokinetic analysis of GSK2982772 following 60 mg BID and 60 mg TID dose at indicated time points. The pharmacokinetic analysis was performed using non-compartmental methods. The analysis was based on Pharmacokinetic Population which comprised of participants in the 'Safety' Population for whom a pharmacokinetic sample was obtained and analyzed.
Time Frame: Day 43 (Pre-dose) and Day 85
Population: Pharmacokinetic Population. Only those participants with data available at specified time points were analyzed (represented by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 23 | 24
Nanograms per milliliter
  Pre-dose on Day 43; n=20, 23: number analyzed (Participants) | 20 | 23
  Pre-dose on Day 43; n=20, 23 | 16.905 (11.1855) | 70.422 (113.6397)
  Day 85; n=20, 22: number analyzed (Participants) | 20 | 22
  Day 85; n=20, 22 | 73.928 (160.0059) | 82.694 (152.4812)

12. Secondary Outcome: Post-dose Plasma Concentrations of GSK2982772 on Days 1 and 43
Description: Blood samples were collected for pharmacokinetic analysis of GSK2982772 following 60 mg BID and 60 mg TID dose at indicated time points. The pharmacokinetic analysis was performed using non-compartmental methods.
Time Frame: 1, 2, 4 and 6 Hours Post-dose on Days 1 and 43
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 23 | 24
Nanograms per milliliter
  1 Hour Post-dose; Day 1; n=22, 24: number analyzed (Participants) | 22 | 24
  1 Hour Post-dose; Day 1; n=22, 24 | 702.547 (342.9405) | 681.675 (293.8436)
  2 Hours Post-dose; Day 1; n=22, 24: number analyzed (Participants) | 22 | 24
  2 Hours Post-dose; Day 1; n=22, 24 | 656.409 (244.9217) | 664.417 (198.8327)
  4 Hours Post-dose; Day 1; n=22, 24: number analyzed (Participants) | 22 | 24
  4 Hours Post-dose; Day 1; n=22, 24 | 262.377 (113.1955) | 249.583 (86.0919)
  6 Hours Post-dose; Day 1; n=22, 24: number analyzed (Participants) | 22 | 24
  6 Hours Post-dose; Day 1; n=22, 24 | 135.923 (67.9503) | 176.567 (194.8144)
  1 Hour Post-dose; Day 43; n=20, 23: number analyzed (Participants) | 20 | 23
  1 Hour Post-dose; Day 43; n=20, 23 | 639.420 (355.1716) | 858.261 (391.7822)
  2 Hours Post-dose; Day 43; n=20, 23: number analyzed (Participants) | 20 | 23
  2 Hours Post-dose; Day 43; n=20, 23 | 579.100 (134.6629) | 690.652 (187.1950)
  4 Hours Post-dose; Day 43; n=20, 23: number analyzed (Participants) | 20 | 23
  4 Hours Post-dose; Day 43; n=20, 23 | 309.700 (114.8441) | 304.348 (136.1582)
  6 Hours Post-dose; Day 43; n=20, 23: number analyzed (Participants) | 20 | 23
  6 Hours Post-dose; Day 43; n=20, 23 | 133.550 (68.6742) | 154.809 (124.4455)

13. Secondary Outcome: Adjusted Mean Percentage Change in Histopathological Scoring of Psoriatic Lesional Biopsy Following Administration of GSK2982772
Description: A target lesion for biopsy was identified on the trunk or extremities at indicated time points. The manual cell counting performed on stained tissue section was referred as histopathological scoring of psoriatic lesions. Histologic assessment included measurement of Cluster of differentiation 11 (CD11+), CD161+, CD3+ and Elastase. Baseline is defined as the latest pre-dose assessment. Percentage change from Baseline was determined from the back-calculation of the log ratio to Baseline. Data for all the listed biomarkers from skin biopsy has been presented for two skin types; dermis and epidermis at Day 43. Due to major Baseline imbalances in psoriasis Baseline characteristics between the BID and TID groups, placebo BID and placebo TID arms were reported separately for all biomarker analyses. NA indicates that data was not available as geometric coefficient of variation could not be calculated for single participant.
Time Frame: Baseline (Pre-dose on Day 1) and Day 43
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percent change
Groups:
- Placebo BID: Eligible participants received placebo BID, oral tablet in Cohort 1 of the study for 12 Weeks.
- Placebo TID: Eligible participants received placebo TID, oral tablet in Cohort 2 of the study for 12 Weeks.
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 10 | 8 | 23 | 24
Percent change
  CD11+; Dermis; n=8, 7, 18 ,23: number analyzed (Participants) | 8 | 7 | 18 | 23
  CD11+; Dermis; n=8, 7, 18 ,23 | 0.4 (44.6) | -9.8 (61.9) | -45.5 (127.8) | -46.6 (93.6)
  CD11+; Epidermis; n=4 ,6, 10, 20: number analyzed (Participants) | 4 | 6 | 10 | 20
  CD11+; Epidermis; n=4 ,6, 10, 20 | -29.7 (278.0) | 4.5 (176.8) | -68.2 (191.6) | -31.5 (157.6)
  CD161+; Dermis; n=7, 7, 13, 23: number analyzed (Participants) | 7 | 7 | 13 | 23
  CD161+; Dermis; n=7, 7, 13, 23 | 23.3 (148.2) | -26.9 (49.5) | -10.7 (73.4) | -14.8 (65.7)
  CD161+; CD161+; Epidermis; n=1, 2 ,0, 4: number analyzed (Participants) | 1 | 2 | 0 | 4
  CD161+; CD161+; Epidermis; n=1, 2 ,0, 4 | -96.7 (NA) — NA indicates that data was not available as geometric coefficient of variation could not be calculated for single participant. | -29.3 (52.1) |  | 13.6 (51.0)
  CD3+; Dermis; n=8 ,7, 20, 23: number analyzed (Participants) | 8 | 7 | 20 | 23
  CD3+; Dermis; n=8 ,7, 20, 23 | -6.3 (52.1) | 4.9 (25.8) | -36.2 (102.3) | -26.0 (57.9)
  CD3+; Epidermis; n=8, 7, 20, 23: number analyzed (Participants) | 8 | 7 | 20 | 23
  CD3+; Epidermis; n=8, 7, 20, 23 | 51.3 (68.9) | 87.8 (48.5) | -40.9 (120.5) | -33.6 (76.0)
  Elastase; Dermis; n=6, 5, 17, 19: number analyzed (Participants) | 6 | 5 | 17 | 19
  Elastase; Dermis; n=6, 5, 17, 19 | -23.3 (46.1) | -50.0 (96.4) | -51.8 (778.4) | -67.4 (527.3)
  Elastase; Epidermis; n=4, 4, 4, 9: number analyzed (Participants) | 4 | 4 | 4 | 9
  Elastase; Epidermis; n=4, 4, 4, 9 | -27.3 (272.2) | -60.8 (177.8) | -36.6 (127.1) | -63.1 (127.5)

14. Secondary Outcome: Adjusted Mean Percentage Change in Histopathological Scoring of Psoriatic Lesional Biopsy: Epidermis Thickness
Description: A target lesion for biopsy was identified on the trunk or extremities at indicated time points. The manual cell counting performed on stained tissue section was referred as histopathological scoring of psoriatic lesions. Histologic assessment included measurement of epidermis thickness. Baseline is defined as the latest pre-dose assessment. Percentage change from Baseline was determined from the back-calculation of the log ratio to Baseline. Due to major Baseline imbalances in psoriasis Baseline characteristics between the BID and TID groups, placebo BID and placebo TID arms were reported separately for all biomarker analyses.
Time Frame: Baseline (Pre-dose on Day 1) and Day 43
Population: Safety Population. Only those participants with data available at specified time point were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percent change
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 8 | 7 | 20 | 23
Percent change | -0.8 (36.4) | -5.7 (25.7) | -22.9 (46.4) | -30.0 (46.0)

15. Secondary Outcome: Number of Participants With Changes in Keratin 16 (K16) Histopathological Scoring in Psoriatic Lesional Biopsies
Description: A target lesion for biopsy was identified on the trunk or extremities at indicated time points. The manual cell counting performed on stained tissue section was referred as histopathological scoring of psoriatic lesions. Histologic assessment included measurement of K16 as keratin expression. Baseline is defined as the latest pre-dose assessment. Results for K16 were categorized as, negative to positive, no change and positive to negative at Day 43. Due to major Baseline imbalances in psoriasis Baseline characteristics between the BID and TID groups, placebo BID and placebo TID arms were reported separately for all biomarker analyses.
Time Frame: Baseline (Pre-dose on Day 1) and Day 43
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 10 | 8 | 23 | 24
Participants
  Negative to positive | 0 | 0 | 2 | 0
  No change | 7 | 6 | 14 | 13
  Positive to negative | 1 | 1 | 4 | 10
  Data missing | 2 | 1 | 3 | 1

16. Secondary Outcome: Messenger Ribonucleic Acid (mRNA) Expression of Inflammatory Gene Transcripts in Psoriatic Lesional Biopsies Following Administration of GSK2982772
Description: A target lesion for biopsy was identified on the trunk or extremities at indicated time points. mRNA expression of inflammatory markers and tissue healing were assessed. Data has been presented for inflammatory gene transcripts including interferon gamma, interleukin 10, interleukin 17A, interleukin 21, interleukin 22, interleukin 23 subunit alpha, interleukin 4 and tumor necrosis factor. Due to major Baseline imbalances in psoriasis Baseline characteristics between the BID and TID groups, placebo BID and placebo TID arms were reported separately for all biomarker analyses.
Time Frame: Day 1 and Day 43
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Copies per 25 nanogram RNA
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 10 | 8 | 23 | 24
Copies per 25 nanogram RNA
  Interferon gamma; Day 1; n=10,8,22,24: number analyzed (Participants) | 10 | 8 | 22 | 24
  Interferon gamma; Day 1; n=10,8,22,24 | 7535938.32 (73.9) | 7224169.85 (82.4) | 6855132.73 (82.4) | 7502338.81 (56.9)
  Interferon gamma; Day 43; n=8, 7, 21, 22: number analyzed (Participants) | 8 | 7 | 21 | 22
  Interferon gamma; Day 43; n=8, 7, 21, 22 | 7467009.88 (91.5) | 5426422.73 (76.7) | 8560810.28 (86.9) | 10082945.49 (73.9)
  Interleukin 10; Day 1; n=10,8,22,24: number analyzed (Participants) | 10 | 8 | 22 | 24
  Interleukin 10; Day 1; n=10,8,22,24 | 5999323.22 (53.3) | 11016442.52 (25.4) | 6319300.05 (49.7) | 9202484.60 (58.2)
  Interleukin 10; Day 43; n=8, 7, 21, 22: number analyzed (Participants) | 8 | 7 | 21 | 22
  Interleukin 10; Day 43; n=8, 7, 21, 22 | 5443660.53 (69.8) | 8948437.47 (37.2) | 6171220.22 (55.7) | 10536204.86 (59.4)
  Interleukin 17A; Day 1; n=10,8,22,24: number analyzed (Participants) | 10 | 8 | 22 | 24
  Interleukin 17A; Day 1; n=10,8,22,24 | 10934904.83 (168.5) | 6066981.63 (247.0) | 7124531.63 (123.0) | 9464750.94 (65.8)
  Interleukin 17A; Day 43; n=8, 7, 21, 22: number analyzed (Participants) | 8 | 7 | 21 | 22
  Interleukin 17A; Day 43; n=8, 7, 21, 22 | 9978712.02 (135.3) | 3694360.37 (311.7) | 6506580.40 (141.8) | 9161452.47 (203.6)
  Interleukin 21; Day 1; n=10,8,22,24: number analyzed (Participants) | 10 | 8 | 22 | 24
  Interleukin 21; Day 1; n=10,8,22,24 | 1947669.71 (129.0) | 1603798.85 (163.3) | 1284591.79 (109.9) | 1210894.24 (93.1)
  Interleukin 21; Day 43; n=8, 7, 20, 22: number analyzed (Participants) | 8 | 7 | 20 | 22
  Interleukin 21; Day 43; n=8, 7, 20, 22 | 1401657.00 (125.0) | 1082550.27 (133.2) | 1215077.05 (106.4) | 1425030.28 (153.4)
  Interleukin 22; Day 1; n=10,8,22,24: number analyzed (Participants) | 10 | 8 | 22 | 24
  Interleukin 22; Day 1; n=10,8,22,24 | 6561087.14 (239.1) | 3042893.44 (191.1) | 3365114.12 (179.5) | 4229367.55 (81.0)
  Interleukin 22; Day 43; n=8, 7, 21, 22: number analyzed (Participants) | 8 | 7 | 21 | 22
  Interleukin 22; Day 43; n=8, 7, 21, 22 | 8431498.86 (125.0) | 1447903.44 (524.1) | 2845767.51 (158.3) | 3457287.68 (200.4)
  Interleukin 23 subunit alpha; Day 1; n=10,8,22,24: number analyzed (Participants) | 10 | 8 | 22 | 24
  Interleukin 23 subunit alpha; Day 1; n=10,8,22,24 | 8747667.18 (131.1) | 6133986.57 (58.2) | 6380211.10 (47.4) | 7006520.16 (56.9)
  Interleukin 23 subunit alpha; Day 43; n=8,7,21,22: number analyzed (Participants) | 8 | 7 | 21 | 22
  Interleukin 23 subunit alpha; Day 43; n=8,7,21,22 | 8552003.39 (91.5) | 5420509.57 (104.6) | 7441092.54 (94.7) | 8918350.71 (82.4)
  Interleukin 4; Day 1; n=10,8,22,24: number analyzed (Participants) | 10 | 8 | 22 | 24
  Interleukin 4; Day 1; n=10,8,22,24 | 461551.13 (131.1) | 596608.00 (102.9) | 800420.91 (62.0) | 514256.12 (75.3)
  Interleukin 4; Day 43; n=7, 7, 21, 22: number analyzed (Participants) | 7 | 7 | 21 | 22
  Interleukin 4; Day 43; n=7, 7, 21, 22 | 416943.25 (144.1) | 492015.71 (69.8) | 671471.18 (75.3) | 438086.02 (69.8)
  Tumor necrosis factor; Day 1; n=10,8,22,24: number analyzed (Participants) | 10 | 8 | 22 | 24
  Tumor necrosis factor; Day 1; n=10,8,22,24 | 43877326.09 (38.3) | 63371891.45 (35.0) | 44208132.84 (27.5) | 63817136.53 (42.8)
  Tumor necrosis factor; Day 43; n=8, 7, 21, 22: number analyzed (Participants) | 8 | 7 | 21 | 22
  Tumor necrosis factor; Day 43; n=8, 7, 21, 22 | 53240969.92 (37.2) | 66678436.36 (50.9) | 52197166.80 (50.9) | 82816773.41 (47.4)

17. Secondary Outcome: Percentage Change From Baseline Psoriatic Lesion Severity Sum (PLSS) Scores in the Index Lesion Following Administration of GSK2982772
Description: Two plaques were selected, one for clinical assessment (index plaque) and one for biopsy. Each lesion was evaluated for 3 components: erythema, induration, and scaling. Each component was given a score using a scale ranging from 0 (no symptom) to 4 (very marked) with increasing score reflecting increased lesion severity. The PLSS is the sum of the erythema, scaling and plaque thickness scores. The total PLSS score ranged from 0 (no symptom) to 12 (very marked). Each lesion must have a PLSS score of >=5. Baseline is defined as the latest pre-dose assessment. Percentage change from Baseline was determined from the back-calculation of the log ratio to Baseline. Due to major Baseline imbalances in psoriasis Baseline characteristics between the BID and TID groups, placebo BID and placebo TID arms were reported separately for all efficacy analyses.
Time Frame: Baseline (Pre-dose on Day 1) and Days 15, 29, 43, 57, 71, 85
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 10 | 8 | 23 | 24
Percentage change
  DAY 15; n=10, 7, 22, 24: number analyzed (Participants) | 10 | 7 | 22 | 24
  DAY 15; n=10, 7, 22, 24 | -0.4 (8.68) | -9.6 (15.79) | -6.7 (14.01) | -7.8 (18.05)
  DAY 29; n=9, 7, 22, 24: number analyzed (Participants) | 9 | 7 | 22 | 24
  DAY 29; n=9, 7, 22, 24 | -8.7 (15.84) | -18.7 (20.09) | -14.3 (21.13) | -16.8 (19.77)
  DAY 43; n=9, 7, 21, 23: number analyzed (Participants) | 9 | 7 | 21 | 23
  DAY 43; n=9, 7, 21, 23 | -10.8 (20.52) | -22.6 (24.24) | -20.7 (19.87) | -27.4 (18.08)
  DAY 57; n=8, 6, 21, 22: number analyzed (Participants) | 8 | 6 | 21 | 22
  DAY 57; n=8, 6, 21, 22 | -11.3 (24.41) | -40.6 (9.58) | -25.5 (23.09) | -27.9 (20.35)
  DAY 71; n=7, 7, 21 ,22: number analyzed (Participants) | 7 | 7 | 21 | 22
  DAY 71; n=7, 7, 21 ,22 | -13.3 (21.66) | -36.8 (18.37) | -34.4 (28.24) | -32.5 (21.06)
  DAY 85; n=7, 7, 21 ,22: number analyzed (Participants) | 7 | 7 | 21 | 22
  DAY 85; n=7, 7, 21 ,22 | -20.6 (15.95) | -42.9 (28.36) | -30.4 (22.20) | -32.9 (26.76)

18. Secondary Outcome: Actual PLSS Scores in the Index Psoriatic Lesion Following Administration of GSK2982772
Description: Two plaques were selected one for clinical assessment (index plaque) and one for biopsy. Each lesion was evaluated for 3 components: erythema, induration, and scaling. Each component was given a score using a scale ranging from 0 (no symptom) to 4 (very marked) with increasing score reflecting increased lesion severity. The PLSS is the sum of the erythema, scaling and plaque thickness scores. The total PLSS score ranged from 0 (no symptom) to 12 (very marked). Each lesion must have a PLSS score of >=5. Due to major Baseline imbalances in psoriasis Baseline characteristics between the BID and TID groups, placebo BID and placebo TID arms were reported separately for all efficacy analyses.
Time Frame: Days 1, 15, 29, 43, 57, 71 and 85
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo BID | Placebo TID | GSK2982772 60 mg BID | GSK2982772 60 mg TID
Number analyzed (Participants) | 10 | 8 | 23 | 24
Scores on a scale
  DAY 1; n=10, 8, 23, 24 | 6.9 (1.73) | 8.5 (1.51) | 8.1 (1.62) | 7.5 (1.44)
  DAY 15; n=10, 7, 22, 24: number analyzed (Participants) | 10 | 7 | 22 | 24
  DAY 15; n=10, 7, 22, 24 | 6.8 (1.48) | 7.4 (1.90) | 7.6 (2.11) | 6.8 (1.76)
  DAY 29; n=9, 7, 22, 24: number analyzed (Participants) | 9 | 7 | 22 | 24
  DAY 29; n=9, 7, 22, 24 | 6.3 (1.80) | 6.6 (1.62) | 7.0 (2.30) | 6.2 (1.91)
  DAY 43; n=9, 7, 21, 23: number analyzed (Participants) | 9 | 7 | 21 | 23
  DAY 43; n=9, 7, 21, 23 | 6.1 (1.54) | 6.3 (1.98) | 6.5 (2.16) | 5.3 (1.21)
  DAY 57; n=8, 6, 21, 22: number analyzed (Participants) | 8 | 6 | 21 | 22
  DAY 57; n=8, 6, 21, 22 | 6.3 (1.49) | 4.8 (1.47) | 6.2 (2.40) | 5.2 (1.37)
  DAY 71; n=7, 7, 21, 22: number analyzed (Participants) | 7 | 7 | 21 | 22
  DAY 71; n=7, 7, 21, 22 | 6.6 (2.07) | 5.3 (2.14) | 5.6 (2.71) | 4.8 (1.37)
  DAY 85; n=7 ,7 ,21, 22: number analyzed (Participants) | 7 | 7 | 21 | 22
  DAY 85; n=7 ,7 ,21, 22 | 6.0 (1.53) | 4.9 (2.73) | 5.8 (2.28) | 4.8 (1.92)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-SAEs were collected from the start of study treatment until follow-up (up to Day 116)
Description: SAEs and non-SAEs were reported for the Safety Population.
Arm/Group | Placebo | GSK2982772 60 mg BID | GSK2982772 60 mg TID
All-Cause Mortality (participants affected / at risk) | 0/18 | 1/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/18 | 1/23 | 1/24
Other Adverse Events (participants affected / at risk) | 8/18 | 21/23 | 16/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=18) | GSK2982772 60 mg BID (N=23) | GSK2982772 60 mg TID (N=24)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural hypertension (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=18) | GSK2982772 60 mg BID (N=23) | GSK2982772 60 mg TID (N=24)
Nasopharyngitis (Infections and infestations) | 4 | 7 | 7
Headache (Nervous system disorders) | 4 | 10 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0
Fatigue (General disorders) | 0 | 3 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-04-12): https://cdn.clinicaltrials.gov/large-docs/33/NCT02776033/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-24): https://cdn.clinicaltrials.gov/large-docs/33/NCT02776033/SAP_001.pdf